CLINICAL TRIAL: NCT04144595
Title: Association Between Low Plasma Glucose After Oral Glucose Tolerance Test in Pregnancy With Impaired Fetal Growth
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. med Flavio Hernández Castro, Principal investigator, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: GI19-00006
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Oral Glucose Tolerance Test; Low Birth Weight
Keywords: Glucose Tolerance Test; Low Birth Weight
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low plasma glucose: This group will be formed by women with low plasma glucose: fasting plasma glucose (<10th percentile, <65 mg/dL), 1 or 2-hour low plasma glucose results after OGTT.
  Interventions: Diagnostic Test: 2 hour 75 g Oral glucose tolerance test
- Normal plasma glucose: This group will be formed by women with normal plasma glucose: fasting plasma glucose ( ≥10th percentile, ≥65 mg/dL but < 92 mg/dL), 1 or 2-hour normal glucose (< 180 mg/dL and 153 mg/dL, respectively) results after OGTT.
  Interventions: Diagnostic Test: 2 hour 75 g Oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: 2 hour 75 g Oral glucose tolerance test — In pregnant women between 24 and 34 weeks of gestational age, plasma glucose was recorded after an overnight fast. Following consumption of 75 g glucose in 200 mL water over 10 min, the equivalent 1 hour and 2 hour values was recorded

SUMMARY:
Objective: To study the association of low maternal plasma glucose in 2 hour 75 g oral glucose tolerance test (OGTT) in women with impaired birth weight and determinate if this result is predictive of low birth weight (<10th percentile according to the INTERGROWTH-21st newborn weight standards for gestational age/sex).

Materials and methods: OGTT at 24-34 week gestation will be performed in pregnant women, the birth weight will be compared between women with low fasting plasma glucose (FPG) (<10th percentile, <65 mg/dL) and normal FPG (≥10th percentile, ≥ 65 mg/dL) also for 1 and 2-hour plasma glucose (1-h PG/2-h PG). Receiver operating characteristic curve analysis will be used to determine the optimal lower OGTT threshold for the prediction of low birth weight.

DETAILED DESCRIPTION:
Maternal hypoglycemia has been reported to be linked with low birth weight and poor neonatal outcome. OGTT is performed routinely in pregnancy and hypoglycemia following this screening test is often encountered and the implication of this finding for the fetal growth is unclear.

The aim of study will be determinate the association of low maternal plasma glucose in OGTT in women with impaired birth weight and determinate if this result is predictive of low birth weight (<10th percentile according to the INTERGROWTH-21st newborn weight standards for gestational age/sex).

The study population will consist of patients with singleton pregnancies who will undergo OGTT at 24-34 weeks, have regular medical checkups throughout their entire pregnancy, deliver on or after 25 week gestation and fulfill inclusion criteria.

The birth weight will be compared between women with low fasting plasma glucose (FPG) (<10th percentile, <65 mg/dL*) and normal FPG (≥10th percentile, ≥ 65 mg/dL) also for 1 and 2-hour plasma glucose (1-h PG/2-h PG). Receiver operating characteristic curve analysis will be used to determine the optimal lower OGTT threshold for the prediction of low birth weight.

This study will be performed according to the standards of the Helsinki Declaration and approval was obtained from the ethics and educational issues coordinating committee of our University Hospital.

*Determinated previously in a pilot study

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancy who underwent OGTT at 24-34 weeks and had regular medical checkups throughout their entire pregnancy.
* Gestational age was determined based on the last menstrual period. If gestational age according to the last menstrual period differed by more than 7 days from that according to ultrasonography at <11 weeks, the latter was used to assign gestational age.

Exclusion Criteria:

* Inaccurate gestational age
* OGTT being drawn outside the prescribed window of 24 to 34 weeks gestation.
* Patients who could not swallow the OGTT solution or vomited afterward were excluded from the study.
* Patients who were diagnosed with gestational diabetes at any time during their pregnancy were excluded.
* The following comorbidities or complications that could affect fetal growth also were excluded: cardiac disease, preeclampsia, gestational hypertension, tobacco use, alcohol intake, stimulant drugs use, maternal systemic diseases (e.g., hypertension, pregestational diabetes, autoimmune disease, thrombotic disease, thyroid disease), intrauterine infectious diseases (e.g., cytomegalovirus, rubella, toxoplasmosis, syphilis), major neonatal anomalies or genetic and structural disorders (e.g., trisomy 21, trisomy 18, trisomy 13, congenital heart disease), placental disorders, and umbilical cord abnormalities.
* Patients with high risk for preeclampsia, intrauterine growth restriction, trisomy 21, trisomy 18 and trisomy 13 in the first trimester screening test.
* Patients with incomplete or missing data were also excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women at 24-28 week gestation
Study Population: The study population consisted of patients with singleton pregnancies who underwent OGTT at 24-34 weeks, had regular medical checkups throughout their entire pregnancy, had delivered on or after 25 week gestation and had fulfilled inclusion criteria. This study was performed according to the standards of the Helsinki Declaration and approval was obtained from the ethics and educational issues coordinating committee of our University Hospital.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Birth weight <10th percentile | Newborn birth weight delivered on or after 25 week gestation will be recorded within the first hour after delivery
  Birth weight <10th percentile according to the INTERGROWTH-21st newborn weight standards for gestational age/sex.
Birthweight <3th percentile | Newborn birth weight delivered on or after 25 week gestation will be recorded within the first hour after delivery
  Birthweight <3th percentile according to the INTERGROWTH-21st newborn weight standards for gestational age/sex.
Birth weight <2500 g | Newborn birth weight delivered on or after 37 week gestation will be recorded within the first hour after delivery
  Birth weight <2500 g of newborn delivered on or after 37 week gestation

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Hernández Castro, MD PhD, Principal Investigator — Obstetrics Department Universidad Autónoma de Nuevo León
Locations (1):
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nayak AU, Vijay AMA, Indusekhar R, Kalidindi S, Katreddy VM, Varadhan L. Association of hypoglycaemia in screening oral glucose tolerance test in pregnancy with low birth weight fetus. World J Diabetes. 2019 May 15;10(5):304-310. doi: 10.4239/wjd.v10.i5.304. PMID 31139317
- [Result] Shinohara S, Uchida Y, Hirai M, Hirata S, Suzuki K. Relationship between maternal hypoglycaemia and small-for-gestational-age infants according to maternal weight status: a retrospective cohort study in two hospitals. BMJ Open. 2016 Dec 2;6(12):e013749. doi: 10.1136/bmjopen-2016-013749. PMID 27913562
- [Result] Topcu HO, Iskender CT, Celen S, Oskovi A, Uygur D, Erkaya S. Maternal hypoglycemia on 50 g glucose challenge test: outcomes are influenced by fetal gender. J Perinat Med. 2016 May 1;44(4):369-76. doi: 10.1515/jpm-2015-0060. PMID 25918915
- [Result] Rogne T, Jacobsen GW. Association between low blood glucose increase during glucose tolerance tests in pregnancy and impaired fetal growth. Acta Obstet Gynecol Scand. 2014 Nov;93(11):1160-9. doi: 10.1111/aogs.12365. Epub 2014 Mar 26. PMID 24576054
- [Result] Melamed N, Hiersch L, Peled Y, Hod M, Wiznitzer A, Yogev Y. The association between low 50 g glucose challenge test result and fetal growth restriction. J Matern Fetal Neonatal Med. 2013 Jul;26(11):1107-11. doi: 10.3109/14767058.2013.770460. Epub 2013 Feb 27. PMID 23350735
- [Result] Vadakekut ES, McCoy SJ, Payton ME. Association of maternal hypoglycemia with low birth weight and low placental weight: a retrospective investigation. J Am Osteopath Assoc. 2011 Mar;111(3):148-52. PMID 21464263
- [Result] Feinberg JH, Magann EF, Morrison JC, Holman JR, Polizzotto MJ. Does maternal hypoglycemia during screening glucose assessment identify a pregnancy at-risk for adverse perinatal outcome? J Perinatol. 2005 Aug;25(8):509-13. doi: 10.1038/sj.jp.7211336. PMID 15908987
- [Result] Leng J, Hay J, Liu G, Zhang J, Wang J, Liu H, Yang X, Liu J. Small-for-gestational age and its association with maternal blood glucose, body mass index and stature: a perinatal cohort study among Chinese women. BMJ Open. 2016 Sep 15;6(9):e010984. doi: 10.1136/bmjopen-2015-010984. PMID 27633632
- [Derived] Hernandez-Castro F, Berlanga-Garza A, Cruz-Gutierrez MD, Soria-Lopez JA, Villagomez-Martinez GE, Davila-Escamilla IV. Prediction of low birth weight with hypoglycemia in glucose tolerance test. Rev Saude Publica. 2021 May 17;55:30. doi: 10.11606/s1518-8787.2021055002543. eCollection 2021. PMID 34008784